CLINICAL TRIAL: NCT02915900
Title: Method for Determining Optimal FSH Dosage During in Vitro Fertilization (IVF)
Brief Title: Optimising FSH Dosage During in Vitro Fertilization Fertilization (IVF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Peter Zoltan Fedorcsak, Head of Department, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 233978
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Infertility
Keywords: In vitro fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Hormone dosage is calculated by using the new method Gonadotropin removal test.
  Interventions: Other: Gonadotropin removal test
- Routine IVF method (Active Comparator): Hormone dosage is chosen by the clinician according to standard clinical routine.
  Interventions: Other: Routine IVF method

INTERVENTIONS:
Other: Gonadotropin removal test — Patient receives hormone dosage adjusted according to the results of the Gonadotropin removal test.
  Arms: Intervention
Other: Routine IVF method — Patient receives hormone dosage according to the standard dosage regimen, without revealing the results of the Gonadotropin removal test to the clinician.
  Arms: Routine IVF method

SUMMARY:
During in vitro fertilisation (IVF) treatment, women receive hormone stimulation with gonadotropins to induce growth of several ovarian follicles. Selecting the optimal dosage of gonadotropin is important to avoid maturation of too few or too many follicles, which may impair the chances of treatment success, lead to treatment cancellation, or serious side effects.

Motivated by the lack of standardised procedures to estimate the optimal dosage of gonadotropins, a patient-specific test has been developed to predict the optimal hormone dosage. By measuring internalisation of gonadotropin by the patient's monocytes isolated form the peripheral blood ex vivo, the Gonadotropin Removal Test determines whether a patient needs increased or reduced hormon doses.

In this clinical study the investigators compare deviation from optimal outcome at oocyte pick-up day in two patient groups. Optimal outcome of stimulation is defined as 10 oocytes collected in the group of patients matching the inclusion criteria of the study.

The control group receives starting hormone dosage assigned by the clinician according to standard clinical procedures. The intervention group receives starting hormone dosage adjusted according to the results of the Gonadotropin Removal Test.

ELIGIBILITY:
Inclusion Criteria:

* Stimulation according to the mid-luteal phase gonadotropin-releasing hormone-agonist protocol
* Pre-selected starting dose <110 IU or >270 IU FSH

Exclusion Criteria:

* Risk for hyperstimulation
* Polycystic ovary syndrome
* Endometriosis stage >III
* BMI>33
* Anti-mullerian hormone value missing

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Deviation from optimal ovarian response, defined as 10 oocytes collected during transvaginal follicle aspiration | The day of follicle aspiration.
  Difference from optimal ovarian response (defined as 10 oocytes collected) is calculated for each patient. The mean these differences is compared between treatment and control groups.
Consistency of optimal ovarian response during stimulation. | The day of follicle aspiration.
  Difference from optimal ovarian response (defined as 10 oocytes collected) is calculated for each patient. Variance of these differences is compared between treatment and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fedorcsak, MD, PhD, Principal Investigator — OUS-HF
Locations (1):
- Department of Reproductive Medicine, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Data might be shared with patient if requested

REFERENCES:
- See also: patent — https://www.google.com/patents/WO2013132036A1?cl=en